CLINICAL TRIAL: NCT01228162
Title: Influence of Muscle Relaxation With Rocuronium Bromide During General Anaesthesia on Muscle Trauma and Postoperative Analgetic Consumption in Patients With Total Hip Prosthesis Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klinikum Hildesheim GmbH (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Dr. Jens Ebnet, MD, Klinikum Hildesheim GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nr. 5615 Hanover Med. School
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Muscle Relaxation; Muscle Trauma; Analgetic Consumption; Total Hip Replacement
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- general anaesthesia (Experimental): patients receiving general anaesthesia and rocuronium bromide for muscle relaxation
  Interventions: Procedure: effect of muscle relaxation on muscle trauma, control group without relaxation
- spinal anaesthesia (Active Comparator): patients receiving spinal anaesthesia without muscle relaxation
  Interventions: Procedure: effect of muscle relaxation on muscle trauma, control group without relaxation

INTERVENTIONS:
Procedure: effect of muscle relaxation on muscle trauma, control group without relaxation — effect of muscle relaxation on muscle trauma, control group without relaxation

SUMMARY:
The researchers want to investigate the effects of muscle relaxation with rocuronium bromide during general anaesthesia on muscle trauma (serum CK, CRP) and postoperative analgesic consumption in patients with total hip prosthesis replacement (general vs. spinal anaesthesia).

ELIGIBILITY:
Inclusion Criteria:

1. patient agreement
2. indication for total hip replacement
3. age 55 - 80 years
4. weight 65 - 95 kg
5. first intervention
6. ASA classification I - III
7. general and spinal anaesthesia possible in this patient

Exclusion Criteria:

a) neuromuscular diseases b) surgery with muscle trauma (within the last 3 months) c) permanent immobility d) intramuscular injections (within the last 4 weeks) e) medication with opioids f) medication with co-analgetics g) contraindications for general or spinal anaesthesia h) dementia, cognitive dysfunction or sleep apnea

-

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
degree of muscle trauma | 24 hours
  serum CK and CRP levels are measured

SECONDARY OUTCOMES:
consumption of analgetics | 3 days
  consumption of piritramide is measured

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Hildesheim GmbH, Hildesheim, Germany